CLINICAL TRIAL: NCT07092007
Title: Safety and Efficacy Study of NWRD09 in HPV-16 Related Intraepithelial Neoplasia and Cervical Cancer Patients
Brief Title: NWRD09 for HPV-16 Related Intraepithelial Neoplasia and Cervical Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Newish Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NEWISH-HPV-M001
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2024-07

CONDITIONS: Intraepithelial Neoplasia; Cervical Cancer
Keywords: HPV16; Intraepithelial Neoplasia; Cervical Cancer; mRNA vaccine
MeSH Terms: conditions — Carcinoma in Situ; Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: 3+3 dose climb
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A( HPV-16 related Cervical, vaginal, and vulvar intraepithelial neoplasia patients ) (Experimental): Patients will be assigned to three dose groups. Each patient will be administered NWRD09 by intramuscular injection. The Maximum Tolerated Dose of NWRD09 will be determined by the classical 3+3 dose escalation schedule. The number of patients will be ranged from 9 to 18.
  Interventions: Biological: NWRD09 administered by intramuscular injection
- Cohort B(HPV-16 related cervical cancer patients) (Experimental): Patients will be assigned to three dose groups. Each patient will be administered NWRD09 by intramuscular injection. The Maximum Tolerated Dose of NWRD09 will be determined by the classical 3+3 dose escalation schedule. The number of patients will be ranged from 9 to 18.
  Interventions: Biological: NWRD09 administered by intramuscular injection

INTERVENTIONS:
Biological: NWRD09 administered by intramuscular injection — NWRD09 administered by intramuscular injection according to the study protocol.

SUMMARY:
This is a single-arm, open label, two cohorts, multi-center clinical study to evaluate the safety and efficacy of HPV-16 targeted mRNA vaccine (NWRD09) in HPV-16 related Cervical, vaginal, and vulvar intraepithelial neoplasia (LSIL and HSIL) patients (cohort A) and HPV-16 related cervical cancer patients (cohort B).

DETAILED DESCRIPTION:
This study is divided into three dose groups in two cohorts. Each patient will be administered NWRD09 by intramuscular injection. The Maximum Tolerated Dose of NWRD09 will be determined by the classical 3+3 dose escalation schedule. The number of patients will be ranged from 9 to 18.

For cohort A, the subjects shall continue to receive safety follow-up until 14 days after the last administration. Colposcopy and biopsy were performed at week 24.

For cohort B, the subjects shall continue to receive safety follow-up until 14 days after the last administration. Imaging evaluation was performed every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for cohort A:

Patients had to meet all of the following inclusion criteria:

1. Women aged between 18 and 60 years.
2. HPV16 is positive during the screening period.
3. Histologically confirmed HPV-16-associated cervical, vaginal, and vulvar intraepithelial neoplasia (LSIL and HSIL). In the case of LSIL, it is necessary to meet persistent HPV16 infection for more than 6 months. In the case of HSIL, it is necessary to meet the requirements of satisfactory colposcopy at screening, which is defined as the squamous columnar epithelial junction (class I or class II transformation zone) is fully visible, and the upper limit of the white epithelium acetate or suspected CIN lesions are fully visible.
4. Eligible subjects of childbearing potential must agree to use a reliable method of contraception (hormonal or barrier method or abstinence, etc.) with their partner for the duration of the trial or for at least 6 months after the last dose. For premenopausal women with the possibility of childbearing, blood pregnancy tests must be negative within 7 days prior to the first use of the NWRD09.
5. Have fully understood the study and voluntarily signed the ICF, have good communication with the investigator, and are able to complete all treatments, examinations, and visits stipulated in the study protocol.

Inclusion criteria for cohort B:

Patients had to meet all of the following inclusion criteria:

1. Women aged ≥ 18 years.
2. HPV16-related recurrent or metastatic advanced cervical cancer (Histologically confirmed squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma) patients who have progressed after at least one lines of standard therapy or are intolerant to toxic side effects, or for which there is no standard treatment at present (Treatment failure refers to: disease progression during or after treatment with systemic antineoplastic regimens; Intolerance refers to: the patient has grade 3-4 adverse reactions after receiving standard therapy, and the patient refuses to continue the original treatment).
3. At least 1 measurable lesion (RECIST 1.1). Tumor lesions that have received prior radiotherapy or other local therapy are considered measurable only if disease progression at the treatment site is clearly documented after completion of treatment.
4. Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1.
5. Had recovered from all toxicities related to prior anticancer therapies to grade≤1 or baseline level as defined by CTCAE v5.0 (except for the asymptomatic laboratory examination abnormalities such as elevated ALP, hyperuricemia, elevated serum amylase/lipase, elevated blood glucose, etc., and toxicities judged by the investigator to have no safety risk, such as alopecia, grade 2 peripheral neurotoxicity, and hypothyroidism stabilized by hormone replacement therapy, etc.).
6. Major organ functions must meet the following criteria:

   1. Blood routine: absolute neutrophil count (ANC) ≥ 1.5×10^9/L, platelet count ≥ 80×10^9/L, hemoglobin ≥ 90 g/L,
   2. Liver function: total bilirubin (TBIL) ≤ 1.5 ULN (≤ 3 ULN for Gilbert's syndrome, liver cancer, or liver metastases), AST and ALT ≤ 2.5 ULN for subjects without liver metastases, and ≤ 5.0 ULN for subjects with liver metastases,
   3. Renal function: creatinine (Cr) ≤ 1.5 ULN, or creatinine clearance (Ccr) ≥ 50 mL/min (using the Cockcroft and Gault formula),
   4. Coagulation function: international normalized ratio (INR) ≤ 1.5, and activated partial thromboplastin time (APTT) ≤ 1.5 ULN.
7. Has life expectancy of at least 3 months in the best judgement of the investigator.
8. Eligible subjects of childbearing potential must agree to use a reliable method of contraception (hormonal or barrier method or abstinence, etc.) with their partner for the duration of the trial or for at least 6 months after the last dose. For premenopausal women with the possibility of childbearing, blood pregnancy tests must be negative within 7 days prior to the first use of the NWRD09.
9. Have fully understood the study and voluntarily signed the ICF, have good communication with the investigator, and are able to complete all treatments, examinations, and visits stipulated in the study protocol.

Exclusion Criteria:

Exclusion criteria for cohort A:

Patients with any of the following were excluded from the study:

1. Any histopathologically confirmed adenocarcinoma or adenocarcinoma in situ (AIS) or invasive cancer.
2. Pregnant, breastfeeding, or planning to conceive during the study period.
3. Received any non-live vaccine injection within 2 weeks prior to the first dose of NWRD09.
4. Received any live vaccine injection within 4 weeks prior to the first dose of NWRD09.
5. Received treatment for LSIL or HSIL within 4 weeks prior to the first dose of NWRD09.
6. Participated in another clinical trial or is in the observation period of another clinical trial within 30 days prior to screening.
7. Continuous (more than 1 week) use of corticosteroids (equivalent to >10 mg/day of prednisone) within 30 days prior to screening, except for hormone replacement therapy and local administration such as inhaled or ocular treatments.
8. History of immunodeficiency or autoimmune diseases (e.g., rheumatoid arthritis, systemic lupus erythematosus, multiple sclerosis).
9. Current or anticipated use of disease-modifying antirheumatic drugs (e.g., azathioprine, cyclophosphamide, cyclosporine, methotrexate) and biological agents (e.g., infliximab, adalimumab, etanercept).
10. Continuous (more than 1 week) use of immunosuppressants (e.g., cyclosporine, tacrolimus, azathioprine, 6-mercaptopurine, and anti-lymphocyte globulin) within 30 days prior to screening.
11. History of solid organ or bone marrow transplantation.
12. Past or current malignancies, except for adequately treated and completely cured ductal carcinoma in situ of the breast, basal cell carcinoma of the skin, superficial bladder tumors, or any other malignancies cured more than 5 years before entering the study.
13. Uncontrolled severe infections (>Grade 2 NCI-CTCAE adverse events, version 5.0).
14. History of HIV infection or syphilis carrier.
15. Active infection (e.g., acute bacterial infection, tuberculosis, active syphilis, active phase of herpes zoster virus infection, active hepatitis B or C, etc.).

    ① Active hepatitis C is defined as: positive hepatitis C antibody and HCV-RNA positive.

    ② Active HIV infection is defined as: positive HIV antibody.

    ③ Active hepatitis B is defined as: HBV titer ≥ 2000 IU/mL (except for subjects who have received anti-HBV treatment for at least 14 days before the first dose and agree to continue antiviral therapy during the study period).
16. Severe allergy history, or history of atopic diseases, or an allergic constitution, if any of these are met.
17. History of severe or multiple hypersensitivity to drugs or pharmaceutical preparations.
18. History of severe local or systemic reaction to vaccines, defined as:

    1. Local reaction: extensive, indurated redness and swelling involving most of the arm, unresolved within 72 hours.
    2. Systemic reaction: persistent fever ≥ 39.5°C within 48 hours. bronchospasm. laryngeal edema. syncope. convulsions or encephalopathy within 72 hours.
19. Severe dysfunction of other organs or heart and lung diseases.
20. History of definite neurological or psychiatric disorders, including epilepsy or dementia.
21. History of drug abuse or alcoholism.
22. Pregnant or breastfeeding women, or women of childbearing age with a positive blood pregnancy test, or patients and their partners of childbearing potential unwilling to use effective contraception during the clinical study and for 6 months after the end of treatment.
23. Patients deemed unsuitable to participate in this clinical trial by the investigator.

Exclusion criteria for cohort B:

Patients with any of the following were excluded from the study:

1. Cervical carcinoma in situ that can be cured by local treatment or non-HPV related cervical cancer.
2. Has not recovered or be reasonably explained from all toxicities related to prior treatments such as surgery, radiotherapy, chemotherapy, immunotherapy, etc.
3. Participated in another clinical trial or is in the observation period of another clinical trial within 30 days prior to screening.
4. Received any non-live vaccine injection within 2 weeks prior to the first dose.
5. Received any live vaccine injection within 4 weeks prior to the first dose.
6. Continuous (more than 1 week) use of corticosteroids (equivalent to >10 mg/day of prednisone) within 30 days prior to screening, except for hormone replacement therapy and local administration such as inhaled or ocular treatments.
7. History of immunodeficiency or autoimmune diseases (e.g., rheumatoid arthritis, systemic lupus erythematosus, multiple sclerosis).
8. Current or anticipated use of disease-modifying antirheumatic drugs (e.g., azathioprine, cyclophosphamide, cyclosporine, methotrexate) and biological agents (e.g., infliximab, adalimumab, etanercept).
9. Continuous (more than 1 week) use of immunosuppressants (e.g., cyclosporine, tacrolimus, azathioprine, 6-mercaptopurine, and anti-lymphocyte globulin) within 30 days prior to screening.
10. History of solid organ or bone marrow transplantation.
11. Past or current malignancies, except for adequately treated and completely cured ductal carcinoma in situ of the breast, basal cell carcinoma of the skin, superficial bladder tumors, or any other malignancies cured more than 5 years before entering the study.
12. Central nervous system (CNS) metastases and/or carcinomatous meningitis (meningeal metastasis).
13. Clinically significant or recurrent pleural, peritoneal, or pericardial effusion requiring frequent drainage.
14. Uncontrolled severe infections (>Grade 2 NCI-CTCAE adverse events, version 5.0).
15. History of HIV infection or syphilis carrier.
16. Active infection (e.g., acute bacterial infection, tuberculosis, active syphilis, active phase of herpes zoster virus infection, active hepatitis B or C, etc.).

    ① Active hepatitis C is defined as: positive hepatitis C antibody and HCV-RNA positive.

    ② Active HIV infection is defined as: positive HIV antibody.

    ③ Active hepatitis B is defined as: HBV titer ≥ 2000 IU/mL (except for subjects who have received anti-HBV treatment for at least 14 days before the first dose and agree to continue antiviral therapy during the study period).
17. Severe allergy history, or history of atopic diseases, or an allergic constitution, if any of these are met.
18. History of severe or multiple hypersensitivity to drugs or pharmaceutical preparations.
19. History of severe local or systemic reaction to vaccines, defined as:

    1. Local reaction: extensive, indurated redness and swelling involving most of the arm, unresolved within 72 hours.
    2. Systemic reaction: fever ≥ 39.5°C within 48 hours. bronchospasm. laryngeal edema. syncope. convulsions or encephalopathy within 72 hours.
20. Severe dysfunction of other organs or heart and lung diseases.
21. History of definite neurological or psychiatric disorders, including epilepsy or dementia.
22. History of drug abuse or alcoholism.
23. Pregnant or breastfeeding women, or women of childbearing age with a positive blood pregnancy test, or patients and their partners of childbearing potential unwilling to use effective contraception during the clinical study and for 6 months after the end of treatment.
24. Patients deemed unsuitable to participate in this clinical trial by the investigator.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 18 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety（Cohort A and B） | From first administration of NWRD09 to 14 days after the last administration
  All adverse events (AE) will be determined based on the rate and severity grade of events, including incidence and severity of serious adverse events (SAE) (according to NCI-CTCAE Standard version 5.0 of common Terms for Adverse Events).
Dose-limiting toxicity (DLT) （Cohort A and B） | 14 days after the first administration
  It would be determined based on the rate and severity grade of events or abnormalities through evaluating systemic or local adverse events, clinical laboratory test results, vital signs that is definitely, probably, or possibly related to the test drug occurring within 21 days of the first dosing will be classified as DLT during dosing climb.

SECONDARY OUTCOMES:
Immunogenicity （Cohort A and B） | To week 24.
  Immunologic reactogenicity by measuring HPV16 E6/E7 specific T cell response (IFN-γ ELISPOT) in blood samples.
Histopathology outcome and HPV Viral clearance （Cohort A） | To week 24.
  Number of subjects with virologically-proven clearance of HPV 16 and number of subjects with histopathological regression of cervical lesions to CIN 1 or normal.
Objective Response Rate (ORR) （Cohort B） | To week 24.
  bjective Response Rate (ORR), defined as the proportion of patients who have either confirmed CR or confirmed PR as best overall response per RECIST 1.1.
Progression-free survival (PFS) （Cohort B） | To week 24.
  Progression-free survival (PFS), defined as the time from the NWRD09 treatment start date to the date of the first documented progression or death from any cause, whichever occurs first.
Duration of response (DOR) （Cohort B） | To week 24.
  Duration of response (DOR), defined as time from the date of first documented response of CR or PR to the date of the first documented progression or death due to any cause.
Disease control rate (DCR) （Cohort B） | To week 24.
  Disease control rate (DCR), defined as is the percentage of evaluable cases with response (PR + CR) and stable disease (SD) after treatment, DCR = CR + PR + SD.

CONTACTS AND LOCATIONS:
Locations (1):
- Heze Municipal Hospita, Heze, Shandong, China

IPD SHARING:
Plan to Share IPD: No